CLINICAL TRIAL: NCT05669820
Title: Antisecretory Factor During Concomitant and Adjuvant Therapy of Primary Glioblastoma, a Randomised, Prospective and Double Blinded Study
Brief Title: Antisecretory Factor Glioblastoma Phase 2
Acronym: AFGB2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peter Siesjö (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FPAFGB2ver6
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: Antisecretory factor; Trials, Randomized Clinical
MeSH Terms: conditions — Glioblastoma | interventions — antisecretory factor

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eggyolk powder with same smell, texture and colour in identical packages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salovum (Active Comparator): Salovum, an egg yolk powder will be orally at dose of 11 g 3 times daily.
  Interventions: Dietary Supplement: Salovum
- Placebo (Placebo Comparator): Placebo, an egg yolk powder will be orally at dose of 11 g 3 times daily.
  Interventions: Dietary Supplement: Placebo egg yolk powder

INTERVENTIONS:
Dietary Supplement: Salovum — Salovum is an eggyolkpowder derived from hens fed with SPC (specially processed cereals) and contains increased amounts of the endogenous protein antisecretory factor.
  Other Names: Antisecretory factor
  Arms: Salovum
Dietary Supplement: Placebo egg yolk powder — Egg yolk powder derived from hen fed with normal feed.
  Arms: Placebo

SUMMARY:
This is a randomised, double blinded and multiple center , Phase 2 study in patients with newly diagnosed glioblastoma. Participants will receive an egg powder enriched for antisecretory factor (AF), Salovum, or a placebo egg powder daily from 2 days before concomitant radio-chemo therapy or chemotherapy until 14 days after finalisation plus during adjuvant chemotherapy.The primary aims of are overall survival at 6 and 12 months after diagnosis

DETAILED DESCRIPTION:
Glioblastoma (GB) is the most common primary brain tumor and also has the worst prognosis with a mean survival time below 1 year and a 5-year survival rate of less than 2%. AF is a 41kilodalton endogenous and essential protein with antisecretory and anti-inflammatory effects. Endogenous AF activity increases after exposure to bacterial toxins and endogenous triggers of inflammation. The active amino-terminal portion of AF has been synthesized as a 16 amino acid peptide (AF-16) and has been used in animal experimental studies. Salovum® is a product based on egg yolk powder B221® and contains high levels of AF. Salovum® is classified as food for special medicinal purposes (FSMP) by the European Union an din other countries.

Many tumors show elevated interstitial fluid pressure (IFP) compared to the surrounding tissue due to vascular leakage, providing a barrier for drug uptake in solid tumors, as well as poor perfusion, resulting in hypoxia and relative resistance to radiochemotherapy.

AF-16 was reported to significantly reduce the IFP in xenotransplanted human glioblastoma by inhibiting an ionic pump, NKCC1, in the tumor tissue. Both Salovum® and AF-inducing specific processed cereals (SPC) prolonged survival in the same models. Systemic temozolomide treatment combined with AF inducing SPC completely blocked tumor growth in GBM xenografts. Likewise, SPC treatment abrogated 90% of pre-established syngeneic tumors in immune competent animals.

Intratumoral delivery of AF-16 potentiated the effect of intratumoral temozolomide in an experimental model of glioblastoma.

Mechanistically, it remains unclear whether AF's effect in tumor models is mediated through decrease of IFP and/or immunomodulation. Also, an effect on the complement system through modulation of circulating complement complexes with proteasome units has been proposed.

Salovum® has been administered to patients with various diseases as, inflammatory bowel disease, Mb Ménière and mastitis and traumatic brain injury without signs of any adverse effects.

In a completed phase1-2 trial in participants with primary gliobalstoma the add on of Salovum during concomitant radiochemotherapa was considered safe and feasible.

The current study is aimed at assessing the efficacy of Salovum in a RCT (randomised controlled trail).

ELIGIBILITY:
Inclusion Criteria:

1. Pathology verified glioblastoma or astrocytoma grade 4
2. Age 18-75 years
3. Surgical treatment-resection.
4. Scheduled concomitant radiochemotherapy, or only chemotherapy.
5. Informed consent

Exclusion Criteria:

1. No informed consent
2. Egg yolk allergy
3. Only surgical biopsy
4. Only radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 12 months from primary surgery
  Survival

SECONDARY OUTCOMES:
Progress free survival at 6 and 12 months | At 6 and 12 months from primary surgery
  Progress free survival as a compound assessment by a multidisciplinary conference (MDC)

OTHER OUTCOMES:
Cognitive function | up to 1 year
  Assessed by Montreal Cognitive Assessment (MoCA)
Neurological function | up to 1 year
  Assessed by Neurologic Assessment in Neuro-Oncology (NANO) scale
QOL Assessed by European Organization of Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C30 | up to 1 years
  Assessed by European Organization of Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) C30 questionnaire
quality of life (QOL) assessed by brain cancer module (BN20) questionnaire | up to 1 years
  Assessed by brain cancer module (BN20) questionnaire
Performance Assessed by Eastern Oncology Cooperative Group (ECOG) performance scale | up to 1 year
  Assessed by Eastern Oncology Cooperative Group (ECOG) performance scale

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Edwardsson, Study Chair — Skane University Hospital; Erik Ehinger, MD, Study Chair — Skane University Hospital
Locations (1):
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
The datasets used and analysed in the current trial will be available in anonymized form after completion of the study, on reasonable request.

REFERENCES:
- [Derived] Ehinger E, Darabi A, Visse E, Edvardsson C, Tomasevic G, Cederberg D, Kinhult S, Rydelius A, Nilsson C, Belting M, Bengzon J, Siesjo P. Antisecretory factor as add-on treatment for newly diagnosed glioblastoma, IDH wildtype: study protocol for a randomized double-blind placebo-controlled trial. Trials. 2025 Mar 13;26(1):86. doi: 10.1186/s13063-025-08792-z. PMID 40083039